CLINICAL TRIAL: NCT02382783
Title: Optimization of the Flare Management in Rheumatoid Arthritis (RA) by Implementing Patient-driven Systematic Changes to the RA Ambulatory Care Stream
Brief Title: Optimizing the Management of Flares in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, John M. Davis, III, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-008535
Record Dates: First submitted 2015-02-23; First posted 2015-03-09 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Disease Activity; Flare; Management of Flares; Pfizer
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FLARE Intervention Group (Other): In the FLARE Intervention Group, we ask that you participate in all of the following, over the course of two years:
  * Baseline Study Visit
  * Monthly: Complete FLARE Questionnaires, at home, and report results. The last question on this questionnaire will ask you if you feel you are having a flare of your disease.
  * FLARE Study Visit (if applicable): We will schedule you to be seen when/if you feel you are having a flare of your disease.
  * Follow-up Visits (minimum of every 6 months): These are done as the standard of care for your RA.
  * At one time-point, during your first return visit after the baseline visit you will have an examination by ultrasound
  * Patient Satisfaction Surveys at three time-points: Baseline, 1 year, 2 year
  Also, your rheumatology health care provider (RHCP) will be asked to participate in the study by completing three satisfaction surveys over the course of two years.
  Interventions: Other: FLARE Intervention Group
- Standard of Care (SOC) Group (No Intervention): If you are randomized to the SOC Group, your care will not be any different than your usual care of rheumatoid arthritis (RA). You will be seen by a rheumatologist at a minimum of every six months, which is the standard of care for RA.
  Additionally (for research), we ask the following of you...
  * At one time-point, during your first return visit after the baseline visit you will have an examination by ultrasound
  * Patient Satisfaction Surveys at three time-points: Baseline, 1 year, 2 year
  Also, your rheumatology health care provider (RHCP) will be asked to participate in the study by completing three satisfaction surveys over the course of two years.

INTERVENTIONS:
Other: FLARE Intervention Group — Everything being completed in this group is also being completed in the Standard of Care (SOC) Group except for the following...
  The participants randomized to this group will be asked to complete FLARE Questionnaires on a monthly basis and will call us each month with their results. The last question on the questionnaire asks if the patient feels he/she is having a flare. If the patient says "yes" to this question, then the study coordinator will arrange for an appointment to be scheduled with a rheumatology health care provider at Mayo Clinic Rochester. The goal will be to have this appointment take place within seven days of the FLARE Questionnaire results being reported.
  Arms: FLARE Intervention Group

SUMMARY:
The purpose of this study is to determine how best to monitor for flares in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This project is aimed at developing an improved multilevel care process model for the management of rheumatoid arthritis (RA) disease activity by implementing systematic self-monitoring of flare experiences by RA patients, combined with continuous patient-tailored adjustments of treatment modalities by a coordinated team of rheumatology health care providers (RHCPs).

ELIGIBILITY:
Inclusion Criteria

* Patient must be ≥ 18 years of age.
* Patient must have been seen by a rheumatology health care provider at least two times within the last 18 months at Mayo Clinic Rochester.
* Patient must have rheumatoid arthritis (RA) according to the 2010 ACR/EULAR classification criteria.
* Patient must have the ability to understand and the willingness to sign a written informed consent document.
* Patient must be willing to return to Mayo Clinic Rochester for follow-up appointments and fill out questionnaires as outlined in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2015-03; Primary Completion 2018-02 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Flare Occurrence | Anticipated length of study is two years.
  The occurrence of flares over the follow-up time (flare rate). The Outcome Measures in Rheumatology(OMERACT-9) definition of flare will be applied to both groups to determine how many occurrences indicate worsening of disease activity, leading to initiation, change, or increase of therapy by RHCPs. This definition will allow for parallel comparisons of flare rates in both groups.
Flare-to-visit Time | Anticipated length of study is two years.
  The flare-to-visit time will be compared between the two groups.

SECONDARY OUTCOMES:
Participant Satisfaction | Three time-points: baseline, year one, and end of study. Anticipated length of study is two years.
  Satisfaction surveys will be provided to participants at three time-points: baseline, year one, and end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Matteson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Bingham CO 3rd, Pohl C, Woodworth TG, Hewlett SE, May JE, Rahman MU, Witter JP, Furst DE, Strand CV, Boers M, Alten RE. Developing a standardized definition for disease "flare" in rheumatoid arthritis (OMERACT 9 Special Interest Group). J Rheumatol. 2009 Oct;36(10):2335-41. doi: 10.3899/jrheum.090369. Epub 2009 Aug 14. PMID 19684147
- [Derived] Myasoedova E, Crowson CS, Giblon RE, McCarthy-Fruin K, Schaffer DE, Wright K, Matteson EL, Davis JM 3rd. Optimization of flare management in patients with rheumatoid arthritis: results of a randomized controlled trial. Clin Rheumatol. 2019 Nov;38(11):3025-3032. doi: 10.1007/s10067-019-04664-5. Epub 2019 Jul 1. PMID 31264032
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials